CLINICAL TRIAL: NCT04736446
Title: Continuous Manual Chest Compressions With Asynchronous Ventilations Using the I-gel Device Versus 30:2 Current Practice Approach With Face Mask Ventilations During Simulated OHCA: Manikin Multicentre Randomised Controlled Trial
Brief Title: Continuous Compressions With Asynchronous Ventilations Using I-gel Device Versus 30:2 Approach During Simulated OHCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geneve TEAM Ambulances (Other)
Collaborators: Service de protection et sauvetage Lausanne (SPSL), Emergency Medical Services, Switzerland (Unknown); Ambulance Riviera, Emergency Medical Services, La Tour-de-Peilz, Switzerland (Unknown); Compagnie d'Ambulances de l'Hôpital du Valais, Emergency Medical Services, Martigny, Switzerland (Unknown); Swissrescue.ch, Website for Prehospital Healthcare Providers, Les Pontins, Switzerland (Unknown); ESAMB - College of Higher Education in Ambulance Care, Geneva, Switzerland (Unknown); STAR Ambulances, Emergency Medical Services, Épalinges, Vaud (Unknown)
Responsible Party: Principal Investigator, Stuby Loric, Paramedic with Certificate of Advanced Studies in Patient Oriented Clinical Research, Geneve TEAM Ambulances
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPR-1
Record Dates: First submitted 2021-01-08; First posted 2021-02-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest; Emergency Medical Services; Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: During pre-scenario sessions (device workshop and 20-minute self-training session) the teams will not have been allocated to one of the study paths.
  Allocation will be discovered as late as possible (after manikin's and defibrillatory characteristics presentation as well as the simulated patient's condition is given). From the moment of the allocation, it will be no more contact between investigators and participants. Due to the nature of the study with us of a supraglottic device, we are not able to blind participants, however they will be unaware of study outcomes. Assessment bias will be limited by using a high-fidelity manikin (SimMan 3G, Laerdal®, Stavanger, Norway) to collect study outcomes. Data analyst will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-gel® group (Experimental): Continuous chest compressions from the start of the CPR with early i-gel® device insertion and asynchronous ventilations
  Interventions: Device: I-gel® supraglottic device
- Standard group (Other): Basic (standard) management by using a ratio of 30 compressions and 2 face mask ventilations
  Interventions: Device: Face mask ventilation

INTERVENTIONS:
Device: I-gel® supraglottic device — Use of an i-gel® supraglottic device to deliver ventilations
  Arms: I-gel® group
Device: Face mask ventilation — Use of a face mask to deliver ventilations
  Arms: Standard group

SUMMARY:
Paramedics and EMT will be recruited among four Emergency Medical Services (EMS) in Switzerland to manage a 10-minutes simulation-based adult out-of-hospital cardiac arrest scenario in teams of two. Depending on randomization, each team will manage the scenario according either to their current approach (30 compressions with 2 bag-mask ventilations), or to the experimental approach (continuous compressions since the start of CPR except for rhythm analysis and shock delivering, with early insertion of an i-gel® device to deliver asynchronous ventilations). The main hypothesis is that early insertion of i-gel could improve CCF during out-of-hospital cardiac arrest, with a reasonable time to first effective ventilation.

DETAILED DESCRIPTION:
Pre-scenario standardized workshop:

First, information about the study will be given and participants' questions are answered. Written consent will be obtained and the first part of the questionnaire individually completed. Participants will be told that the resuscitation scenario will be stopped after 10 minutes, independently of their actions and that no feedback will be given.

Then, the use of i-gel® device use will be taught by one of the investigators (LSt) in accordance with Peyton's approach because this approach has shown superiority, and based on a standard operating procedure created by study investigators following manufacturer's instructions:

1. The instructor performs a complete insertion sequence in real-time without any comments;
2. The instructor performs an insertion sequence with step-by-step explanations (description of key points);
3. The learners guide the instructor step by step to perform the insertion;
4. The learners do the complete insertion sequence then feedback could be given. They will perform this step a maximum of 3 times.

This workshop will last 20 minutes.

Self-managed training session:

After the workshop, each team will have 20 minutes to self-train the introduction of the device in the complete OHCA management sequence on a CPR manikin permitting airway management. They will be supported by a demonstration video, which they could use freely.

Resuscitation scenario:

When entering the study room, an overview of the characteristics of the simulation manikin and the use of the defibrillator will be given through a standardized video. The team will then be asked to perform a 10-minutes highly realistic adult CPR scenario on a high-fidelity WiFi manikin. The procedure will be standardized across all sites to ensure that each participant is exposed to exactly the same case, with similar challenges in decision-making and treatment provided on the same manikin. The uniform delivery of the scenario throughout the entire study will minimize confounders. The room will be exclusively devoted to the simulation to prevent unexpected interruptions or external stimuli.

The scenario will start with a clinical statement to recognize the life-threatening condition of the patient, given by one of the investigators as follows: " Here is Michael, a 50-years old who suddenly collapsed 10 minutes ago. He is now unconscious, pale and seems not breathing. The medical reinforcement is already underway and will be on site in about ten minutes. No first responder were dispatched to the scene and there is no bystander ". The team leader will be asked to reformulate this statement (closed-loop communication) to ensure comprehension. He will then open the following envelope of the stack. The opaque, sealed envelope will contain the approach they will have to apply: standard care or experimental approach. From this point on, there will be no more contact between the participants and the study team, except to stop the scenario.

If the participant checks the breathing, the patient will be apneic and pulse will be absent if checked. The first compression will be defined as T0. After placement of the pads, the defibrillator's display will show ventricular fibrillation (VF). All following rhythm analyses will show refractory VF, regardless of whether a shock is delivered. To increase simulation's fidelity, CPR waves will be displayed when compressions will be delivered. Participants will be able to obtain an intravenous access on first attempt. They should administer first 1 mg of epinephrine (at the earliest after the second shock), then a first-dose of amiodarone or lidocaine following local protocols (in accordance with the 2020 AHA cardiac arrest algorithm. The scenario will be stopped exactly 10 minutes after the first compression. There will be no feedback after the study period.

ELIGIBILITY:
Inclusion Criteria:

* To be a registered paramedic or EMT
* To have previously completed the 20-minute workshop on how using the device by on of the study investigators
* To have previously completed the 20-minute self-training session following a video recorded by the study investigators
* Participation agreement

Exclusion Criteria:

* Member of the study investigators
* To have not undergone the 20-minute workshop
* To have not watch the video

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Chest compressions fraction (CCF) over the first 2 minutes of CPR | At the end of Cycle 1 (each cycle is 2 minutes)
  Proportion of time where compressions are performed during the first two minutes of the scenario

SECONDARY OUTCOMES:
CCF of second cycle | At the end of Cycle 2 (each cycle is 2 minutes)
  Proportion of time where compressions are performed during the following two minutes of the scenario
CCF of third cycle | At the end of Cycle 3 (each cycle is 2 minutes)
  Proportion of time where compressions are performed during the following two minutes of the scenario
CCF of fourth cycle | At the end of Cycle 4 (each cycle is 2 minutes)
  Proportion of time where compressions are performed during the following two minutes of the scenario
CCF of fifth cycle | At the end of Cycle 5 (each cycle is 2 minutes)
  Proportion of time where compressions are performed during the following two minutes of the scenario
Overall CCF | 10 minutes of scenario
  Proportion of time where compressions are performed during the entire scenario
Chest compressions depth | 10 minutes of scenario
  Mean depth of compressions
Proportions of compressions above, below and in the depth target | 10 minutes of scenario
  The depth target is 5 to 6 cm
Chest compressions frequency | 10 minutes of scenario
  Mean frequency of compressions
Proportions of compressions above, below and in the frequency target | 10 minutes of scenario
  The frequency target is 100 to 120 compressions by minute
Time to first shock | 10 minutes of scenario
  Interval between start of compressions and delivering of first shock
Time to first effective ventilation | 10 minutes of scenario
  Interval between start of compressions and delivering of first effective ventilation (defined as volume >300 ml)
Ventilations volume | 10 minutes of scenario
  Mean volume of ventilations
Proportions of ventilations above, below and in the volume target | 10 minutes of scenario
  The volume target is 300 to 700 ml
User satisfaction assessed by a 5-point Likert scale ranging from "Not satisfied" to "Very satisfied" | 10 minutes of scenario
  User satisfaction regarding applied approach assessed on a 5-point Likert scale ranging from "Not satisfied" to "Very satisfied"
Self-assessed cognitive load using a 9-point scale ranging from "Very, very low mentale effort" to "Very, very high mental effort" | 10 minutes of scenario
  Self-reported cognitive load during resuscitation scenario assessed using a 9-point symmetrical category scale which ranged from "Very, very low mental effort" (1) to "Very, very high mental effort" (9),
Chest compression relaxation | 10 minutes of scenario
  Proportion of correct compressions (with less than 5 mm deviation from reference value)
Number of delivered ventilations | 10 minutes of scenario
  Absolute number of delivered ventilations

CONTACTS AND LOCATIONS:
Overall Officials: Loric Stuby, Principal Investigator — Genève TEAM Ambulances
Locations (1):
- Genève TEAM Ambulances, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be deposited on Mendeley Data
Supporting Information: ICF
Time Frame: Starting 6 months after publication for at least two years
Access Criteria: Open access on https://data.mendeley.com/

REFERENCES:
- [Background] Stuby L, Jampen L, Sierro J, Paus E, Spichiger T, Suppan L, Thurre D. Effect on Chest Compression Fraction of Continuous Manual Compressions with Asynchronous Ventilations Using an i-gel(R) versus 30:2 Approach during Simulated Out-of-Hospital Cardiac Arrest: Protocol for a Manikin Multicenter Randomized Controlled Trial. Healthcare (Basel). 2021 Mar 20;9(3):354. doi: 10.3390/healthcare9030354. PMID 33804664
- [Background] Stuby L, Suppan L, Jampen L, Thurre D. Impact of the Over-the-Head Position with a Supraglottic Airway Device on Chest Compression Depth and Rate: A Post Hoc Analysis of a Randomized Controlled Trial. Healthcare (Basel). 2022 Apr 13;10(4):718. doi: 10.3390/healthcare10040718. PMID 35455895
- [Result] Stuby L, Jampen L, Sierro J, Bergeron M, Paus E, Spichiger T, Suppan L, Thurre D. Effect of Early Supraglottic Airway Device Insertion on Chest Compression Fraction during Simulated Out-of-Hospital Cardiac Arrest: Randomised Controlled Trial. J Clin Med. 2021 Dec 31;11(1):217. doi: 10.3390/jcm11010217. PMID 35011958
- See also: Whole project website — https://swiss-cpr-studies.ch/